CLINICAL TRIAL: NCT00282555
Title: Assessment of the Healing Rate of Erosive or Ulcerative Esophagitis After Two and Four Weeks of Treatment With S-Tenatoprazole-Na (STU-Na) 15 mg, 30 mg, 60 mg, 90 mg and Esomeprazole 40 mg. A Multicenter, Randomized, Double-Blind, Parallel Group Study.
Brief Title: Efficiency Study of S-Tenatoprazole-Na to Treat Erosive or Ulcerative Esophagitis
Status: Suspended | Phase: Phase 2 | Type: Interventional
Sponsor: STEBA France (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HEC/STU(-Na)05816N/TU 2.05
Record Dates: First submitted 2006-01-25; First posted 2006-01-26 (Estimated); Last update posted 2008-03-19 (Estimated); Status verified 2008-03

CONDITIONS: Esophagitis, Reflux
Keywords: Esophagitis, Reflux; S-Tenatoprazole-Na; Heartburn; Esophageal endoscopy
MeSH Terms: conditions — Esophagitis, Peptic; Heartburn

INTERVENTIONS:
Drug: S-Tenatoprazole-Na (STU-Na)

SUMMARY:
STU-Na belongs to the proton pump inhibitors (PPI), a group of drugs that reduce gastric acidity. PPI are used to treat acid related diseases like erosive or ulcerative esophagitis. This trial aims to find out the therapeutic dose of STU-Na required for healing patients with erosive or ulcerative esophagitis. One of four dosages of STU-Na (15 mg, 30 mg, 60 mg, or 90 mg daily), or Esomeprazole 40 mg daily, an already marketed PPI, will be given to patients. The attribution to one of the 5 treatment groups will be by chance. Neither the patient nor the study physician will know, which treatment is administered to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients aged 18 to 75 years inclusive
* Symptomatic ulcerative or erosive esophagitis
* Presence of heartburn (daytime and/or nighttime).
* Understanding the study and agreeing to give a written informed consent
* Able to communicate well with the investigator him(her)self or his/her representatives
* Able and agreeing to comply with all study requirements

Exclusion Criteria:

* gastrointestinal bleeding
* gastric or esophageal surgery
* Zollinger-Ellison syndrome
* primary esophageal motility disorders,
* esophageal stricture,
* inflammatory bowel disease,
* upper gastrointestinal malignancy,
* pancreatitis,
* malabsorption
* Barrett's esophagus (> 3 cm)
* Severe disease/condition such as malignancy
* Hypersensitivity to PPIs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450
Dates: Start 2006-02

PRIMARY OUTCOMES:
Esophageal endoscopy: assessment of achievement of grade "not present" in the Los Angeles scale of esophagitis after two weeks of treatment

SECONDARY OUTCOMES:
Esophageal endoscopy: assessment of achievement of grade "not present" in the Los Angeles scale of esophagitis after four weeks of treatment.
Assessment of complete relief of heartburn

CONTACTS AND LOCATIONS:
Overall Officials: Alan Thomson, MD, Prof., Study Chair — University of Alberta, Division of Gastroenterology, Department of Medicine, Edmonton, Alberta, Canada
Locations (17):
- Canada (17):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Abbottsford, British Columbia
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Guelph, Ontario
  - Hamilton, Ontario
  - Scarborough Village, Ontario
  - Toronto, Ontario
  - Windsor, Ontario
  - Lévis, Quebec
  - Montreal, Quebec
  - Pointe-Claire, Quebec
  - Québec, Quebec
  - Sherbrooke, Quebec
  - St-Charles-de-Borromée, Quebec
  - Saskatoon, Saskatchewan

REFERENCES:
- [Background] Armstrong D. Review article: gastric pH -- the most relevant predictor of benefit in reflux disease? Aliment Pharmacol Ther. 2004 Oct;20 Suppl 5:19-26; discussion 38-9. doi: 10.1111/j.1365-2036.2004.02140.x. PMID 15456460
- [Background] Bell NJ, Burget D, Howden CW, Wilkinson J, Hunt RH. Appropriate acid suppression for the management of gastro-oesophageal reflux disease. Digestion. 1992;51 Suppl 1:59-67. doi: 10.1159/000200917. PMID 1397746
- [Background] Burget DW, Chiverton SG, Hunt RH. Is there an optimal degree of acid suppression for healing of duodenal ulcers? A model of the relationship between ulcer healing and acid suppression. Gastroenterology. 1990 Aug;99(2):345-51. doi: 10.1016/0016-5085(90)91015-x. PMID 2142113
- [Background] DeVault KR, Castell DO. Updated guidelines for the diagnosis and treatment of gastroesophageal reflux disease. The Practice Parameters Committee of the American College of Gastroenterology. Am J Gastroenterol. 1999 Jun;94(6):1434-42. doi: 10.1111/j.1572-0241.1999.1123_a.x. No abstract available. PMID 10364004
- [Background] Galmiche JP, Bruley Des Varannes S, Ducrotte P, Sacher-Huvelin S, Vavasseur F, Taccoen A, Fiorentini P, Homerin M. Tenatoprazole, a novel proton pump inhibitor with a prolonged plasma half-life: effects on intragastric pH and comparison with esomeprazole in healthy volunteers. Aliment Pharmacol Ther. 2004 Mar 15;19(6):655-62. doi: 10.1111/j.1365-2036.2004.01893.x. PMID 15023167
- [Background] Horn J. The proton-pump inhibitors: similarities and differences. Clin Ther. 2000 Mar;22(3):266-80; discussion 265. doi: 10.1016/S0149-2918(00)80032-6. PMID 10963283
- [Background] Hunt RH, Armstrong D, James C, Chowdhury SK, Yuan Y, Fiorentini P, Taccoen A, Cohen P. Effect on intragastric pH of a PPI with a prolonged plasma half-life: comparison between tenatoprazole and esomeprazole on the duration of acid suppression in healthy male volunteers. Am J Gastroenterol. 2005 Sep;100(9):1949-56. doi: 10.1111/j.1572-0241.2005.41956.x. PMID 16128938
- [Background] Kakinoki B, Ono C, Yamazaki N, Chikamatsu N, Wakatsuki D, Uchiyama K, Morinaka Y. General pharmacological properties of the new proton pump inhibitor (+/-)-5-methoxy-2-[[(4-methoxy-3,5-dimethylpyrid-2-yl)methyl]sulf inyl]- 1H-imidazo[4,5-b]pyridine. Methods Find Exp Clin Pharmacol. 1999 Apr;21(3):179-87. doi: 10.1358/mf.1999.21.3.534827. PMID 10389120
- [Background] Katz PO, Castell DO, Chen Y, Andersson T, Sostek MB. Intragastric acid suppression and pharmacokinetics of twice-daily esomeprazole: a randomized, three-way crossover study. Aliment Pharmacol Ther. 2004 Aug 15;20(4):399-406. doi: 10.1111/j.1365-2036.2004.02079.x. PMID 15298633
- [Background] Kromer W, Horbach S, Luhmann R. Relative efficacies of gastric proton pump inhibitors: their clinical and pharmacological basis. Pharmacology. 1999 Aug;59(2):57-77. doi: 10.1159/000028306. PMID 10450061
- [Background] Lundell LR, Dent J, Bennett JR, Blum AL, Armstrong D, Galmiche JP, Johnson F, Hongo M, Richter JE, Spechler SJ, Tytgat GN, Wallin L. Endoscopic assessment of oesophagitis: clinical and functional correlates and further validation of the Los Angeles classification. Gut. 1999 Aug;45(2):172-80. doi: 10.1136/gut.45.2.172. PMID 10403727
- [Background] Revicki DA, Crawley JA, Zodet MW, Levine DS, Joelsson BO. Complete resolution of heartburn symptoms and health-related quality of life in patients with gastro-oesophageal reflux disease. Aliment Pharmacol Ther. 1999 Dec;13(12):1621-30. doi: 10.1046/j.1365-2036.1999.00669.x. PMID 10594397
- [Background] Stedman CA, Barclay ML. Review article: comparison of the pharmacokinetics, acid suppression and efficacy of proton pump inhibitors. Aliment Pharmacol Ther. 2000 Aug;14(8):963-78. doi: 10.1046/j.1365-2036.2000.00788.x. PMID 10930890
- [Background] Uchiyama K, Wakatsuki D, Kakinoki B, Takeuchi Y, Araki T, Morinaka Y. The long-lasting effect of TU-199, a novel H+, K(+)-ATPase inhibitor, on gastric acid secretion in dogs. J Pharm Pharmacol. 1999 Apr;51(4):457-64. doi: 10.1211/0022357991772510. PMID 10385219